CLINICAL TRIAL: NCT07214103
Title: Phase IIb Multicenter Randomized Controlled Trial Evaluating the Efficacy of Sivelestat in Patients With Septic Coagulopathy
Acronym: SivelSep
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9415
Record Dates: First submitted 2025-10-02; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Septic Shock; Coagulopathy
MeSH Terms: conditions — Shock, Septic; Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active therapy (Experimental): • Sivelestat
  Interventions: Drug: • Sivelestat intravenous infusion
- Placebo therapy (Placebo Comparator): • NaCl
  Interventions: Drug: NaCl intravenous infusion

INTERVENTIONS:
Drug: • Sivelestat intravenous infusion — * Intervention: Sivelestat 0.20 mg/kg/h via continuous intravenous infusion (IVSE) for 72 hours
  * Anticoagulation: Unfractionated heparin (UFH) at a minimum dose of 100 IU/24h (or higher if required)
  Arms: Active therapy
Drug: NaCl intravenous infusion — * Intervention: NaCl 0.9% (normal saline) via continuous intravenous infusion (IVSE) at the same rate as the experimental group for 72 hours
  * Anticoagulation: Unfractionated heparin (UFH) at a minimum dose of 100 IU/24h (or higher if required)
  Arms: Placebo therapy

SUMMARY:
Sepsis-induced disseminated intravascular coagulation (DIC) is a severe complication occurring in one-third of patients with septic shock, for which no specific treatment currently exists. It results from excessive systemic activation of coagulation and impaired fibrinolysis, leading to the development of disseminated microthromboses. We have recently demonstrated: 1) the contribution of NETs to the hypercoagulability observed in DIC, and 2) the role of neutrophil elastase-bound to NET DNA-in degrading plasminogen, a key factor limiting fibrinolysis and thus preventing the lysis of microthrombi in DIC.

Sivelestat is a neutrophil elastase inhibitor used in Japan for the treatment of acute respiratory distress syndrome (ARDS). It has the potential to inhibit: 1) neutrophil activation and the release of inflammatory mediators, and 2) plasminogen degradation, which drives fibrinolytic failure. A recent meta-analysis including 2,050 patients across 15 studies showed that Sivelestat reduced ARDS patient mortality at day 28-30 (RR = 0.81, 95% CI = 0.66-0.98, p = 0.03), decreased mechanical ventilation duration and ICU length of stay, and improved oxygenation.

We propose to conduct a multicenter, double-blind, placebo-controlled phase IIb trial evaluating the efficacy of Sivelestat in restoring fibrinolysis in patients with septic shock complicated by coagulopathy, defined by a positive SIC score (≥ 4 points).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 85 years
* Patient (male or female) admitted to the ICU with:

  * Septic shock defined by Sepsis-3 criteria: acute, life-threatening organ dysfunction related to a suspected or confirmed infection, requiring vasopressor support to maintain a mean arterial pressure ≥ 65 mmHg and a serum lactate level > 2 mmol/L despite adequate fluid resuscitation.
  * Coagulopathy defined by a SIC score ≥ 4 points.
* Randomization within 12 hours after the diagnosis of coagulopathy (positive SIC score).
* Patient affiliated with a national health insurance system.
* Written informed consent: freely given, dated, and signed.

  * By the patient
  * Or by a legal representative if the patient is unable to provide consent.
  * Or through an emergency inclusion procedure if the patient is unable to consent and no family member is available

Exclusion Criteria:

* History of hypersensitivity reaction to Sivelestat (the only contraindication for Sivelestat)
* Patient weight > 100 kg
* Severe chronic liver disease (Child-Pugh C)
* Contraindication to the use of unfractionated heparin
* Moribund patient at the time of randomization
* Limitation of active therapeutic interventions at the time of study inclusion
* Under legal protection (guardianship, curatorship, or legal safeguard)
* Pregnancy or breastfeeding
* Participation in another interventional drug clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma plasminogen levels | 24 hours
  Change in plasma plasminogen levels after 24 hours of treatment with either placebo or Sivelestat.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France, France